CLINICAL TRIAL: NCT06224751
Title: A Program to Develop Computerised Visual Function Tests for Cross Sectional Routine Clinical Practice and Long Term Monitoring to Detect Adverse Change in Visual Function.
Brief Title: Developing Better Computerised Vision Tests (CVTV)
Acronym: CVTV
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 277317
Record Dates: First submitted 2023-10-25; First posted 2024-01-25 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Visual Impairment; Amblyopia; Macular Degeneration; Ophthalmic Disease
Keywords: Visual acuity; Visual function; Ocular disease
MeSH Terms: conditions — Vision Disorders; Amblyopia; Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Near logMAR letter acuity: Comparison of measurements made with the trial computerised test to the trial gold standard printed test
  Interventions: Diagnostic Test: Near logMAR letter acuity
- Near logMAR word acuity: Comparison of measurements made with the trial computerised test to the trial gold standard printed test
  Interventions: Diagnostic Test: Near LogMAR word acuity
- Letter Contrast Sensitivity: Comparison of measurements made with the trial computerised test to the trial gold standard printed test
  Interventions: Diagnostic Test: Letter Contrast Sensitivity
- Vanishing Optotype Sloan letters: Comparison of measurements made with the trial computerised test to the trial gold standard printed test
  Interventions: Diagnostic Test: Vanishing Optotype Sloan Letters
- Auckland Optotypes/Auckland Vanishing Optotypes: Comparison of measurements made with the trial computerised test to the trial gold standard printed test
  Interventions: Diagnostic Test: Auckland Optotype/Auckland Vanishing Optotypes
- Low contrast letter acuity: Comparison of measurements made with the trial computerised test to the trial gold standard printed test
  Interventions: Diagnostic Test: Low Contrast Letter Acuity
- Red Green Stereoacuity: Comparison of measurements made with the trial computerised test to the trial gold standard printed test
  Interventions: Diagnostic Test: Red Green Stereoacuity

INTERVENTIONS:
Diagnostic Test: Near logMAR letter acuity — Comparison of gold standard printed tests and computerised versions
  Groups: Near logMAR letter acuity
Diagnostic Test: Near LogMAR word acuity — Comparison of gold standard printed tests and computerised versions
  Groups: Near logMAR word acuity
Diagnostic Test: Red Green Stereoacuity — Comparison of gold standard printed tests and computerised versions
  Groups: Red Green Stereoacuity
Diagnostic Test: Auckland Optotype/Auckland Vanishing Optotypes — Comparison of gold standard printed tests and computerised versions
  Groups: Auckland Optotypes/Auckland Vanishing Optotypes
Diagnostic Test: Vanishing Optotype Sloan Letters — Comparison of gold standard printed tests and computerised versions
  Groups: Vanishing Optotype Sloan letters
Diagnostic Test: Letter Contrast Sensitivity — Comparison of gold standard printed tests and computerised versions
  Groups: Letter Contrast Sensitivity
Diagnostic Test: Low Contrast Letter Acuity — Comparison of gold standard printed tests and computerised versions
  Groups: Low contrast letter acuity

SUMMARY:
Clinical vision measurements usually involve printed charts with an eye care professional interpreting patient responses to generate a score. Those scores determine the need for or outcome of treatment. Detecting change can be improved with strict procedures/scoring, lending itself to computerisation. This in turn allows integration with electronic medical records. Many eye tests could be computerised in this way. At Guys and St Thomas' NHS Foundation Trust, the investigators have developed and validated a computerised test of distance visual acuity, called COMPlog which is now in widespread use. The investigators now want to increase the range of tests available.

There is also a need to longitudinally monitor for adverse change. Such monitoring must be developed to keep false positive and false negative change detection to a minimum.

The aims of this two year linked program are to:

Part A) validate an extended range of computerised vision measurement tests against their gold standard hard copy printed equivalents. Some of these tests are designed for use in children and all are meant to quantify both normal and impaired vision. Patients of all ages and visual function will therefore be recruited from St Thomas' Hospital. The specific tests we aim to validate are logMAR Letter Near Acuity, Word Near Acuity, Letter Contrast Sensitivity, Auckland Optotypes Picture Acuity, Low Contrast Letter Acuity, Stereoacuity and Vanishing Optotypes. Patients will undergo test-retest measurements with up to two of these.

Part B) Iteratively develop an application for use in home monitoring of subjects at risk of treatable vision loss due to age related macular degeneration.

All computerised tests in parts A and B will be performed on prototype software. Eye patients will be recruited as subjects. Patients recruited to part A will undergo tests on one day for up to an hour, subjects in part B will participate for between 1 hour and two months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients attending hospital eye clinics, aged 3 - 99, inclusive.
* Patients able to understand the information sheet, and willing and able to give informed consent to participate.
* Patients with visual function ranging from normal to severely impaired.
* Willing and able to comply with the visual function testing protocol.
* Some validation studies require recruitment of disease specific groups (such as children with amblyopia or adults with age related macular degeneration).

For Part B of the project which aims to develop and pilot a home monitoring application, only adult (18-99 years) subjects complying with the above who also own a suitable browser device will be recruited.

Exclusion Criteria:

* Unwilling or unable to comply with the visual function testing protocol.
* Unwilling or unable to give informed consent.
* Unwilling to participate.
* In other research trials.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending the outpatient eye clinics at St Thomas' Hospital NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Test agreement between the computerised vision measurement test and the gold standard hard copy test. | Through study completion, an average of 1 year
  The test agreement is quantified in terms of the mean difference and 95% confidence interval of the mean in log units.
Test-retest variability for the computerised vision measurement test and the gold standard hard copy test. | Through study completion, an average of 1 year
  Measurement variability (difference in two measures captured using the same vision test on the same day) will be quantified in log units for each vision test used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Laidlaw, MD FRCOphth, Principal Investigator — St Thomas' Hospital, London
Locations (1):
- St Thomas' Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No